CLINICAL TRIAL: NCT03039933
Title: Intervention to Reduce Fear of Hypoglycemia and Optimize Type 1 Diabetes Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-0645
Record Dates: First submitted 2016-12-19; First posted 2017-02-01 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Type1diabetes; Fear of Hypoglycemia
MeSH Terms: interventions — Therapeutics; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fear of Hypoglycemia Intervention (Active Comparator): Cognitive behavioral therapy based psychological intervention occurring every other week for 12 weeks.
  Interventions: Behavioral: Fear of Hypoglycemia
- Treatment As Usual (Other): Control group completes questionnaires but does not receive any study intervention. Receives medical care as usual.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: Fear of Hypoglycemia — Participants will receive exposure and response prevention and/or hypoglycemia awareness training.
  Arms: Fear of Hypoglycemia Intervention
Other: Treatment As Usual — Treatment As Usual
  Other Names: Standard of Care
  Arms: Treatment As Usual

SUMMARY:
The overall objective and Primary Aim of this Limited Competition: Small Grant Program (R03) is to address the critical need of identifying and decreasing fear of hypoglycemia, which will be accomplished by conducting a pilot randomized clinical trial to evaluate the efficacy of Blood Glucose Awareness Training, which has been adapted for, but never evaluated in adolescents with Type 1 Diabetes (T1D) and their parents.

ELIGIBILITY:
Inclusion Criteria:

* adolescents aged 10-17 years and their parent(s) or legal guardian;
* T1D duration >1 year;
* insulin pump use >6 months;
* agreement of both parent and adolescent to participate in intervention sessions;
* elevated scores on the Parent Hypoglycemia Fear Survey - Behavior Subscale.

Exclusion Criteria:

* developmental disability or reading disorder that prevents understanding of the intervention materials; and
* non-English speaking adolescents and parents.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Decrease in scores on the Hypoglycemia Fear Survey | Baseline, 3 and 6 months
  To address the critical need of identifying and decreasing fear of hypoglycemia, which will be accomplished by evaluating the efficacy of Blood Glucose Awareness Training as compared to treatment as usual.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Driscoll, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No